CLINICAL TRIAL: NCT04770805
Title: In Utero Fetoscopic Repair Program for Sacral Myelomeningoceles and Mye-LDM
Acronym: PRIUM2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP191101; N° IDRCB: 2020-A01413-36 (Other: ANSM)
Record Dates: First submitted 2021-01-24; First posted 2021-02-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Sacral Myelomeningocele; Neural Tube Defects; Spina Bifida
Keywords: Sacral Myelomeningocele; MyeLDM; Fetal surgery; Fetoscopic Repair Program; Neural Tube Defect; Spina bifida
MeSH Terms: conditions — Neural Tube Defects; Spinal Dysraphism | interventions — Fetoscopy

STUDY DESIGN:
Intervention Model Description: This is a single arm clinical study. All participants will undergo laparotomy with exteriorization of the uterus followed by fetoscopic repair of the fetal MMC/MyeLDM lesion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fetoscopic repair (Experimental): Sacral Myelomeningocele and Mye-LDM Fetoscopic repair
  Interventions: Procedure: Fetoscopy

INTERVENTIONS:
Procedure: Fetoscopy — After an exteriorization of the uterus through a laparotomy, humidified and warmed gas will be insufflated with low pressure (6 to 8mmHg mmHg). Fetoscopic repair surgery will consist in a dissection of the placode, its reintegration into the spinal canal and the closure of the lesion, through a three ports access. After fetal surgery, the gas will be exsufflated and the trocar ports will be closed. The uterus will be reintegrated before suturing the maternal abdominal wall.

SUMMARY:
The purpose of the study is to evaluate the feasibility and the maternal, fetal and postnatal outcomes of sacral myelomeningocele (MMC) and Myelic Limited Dorsal Myeloschisis (MyeLDM) fetoscopic repair at Trousseau Hospital (Paris, France).

DETAILED DESCRIPTION:
Myelomeningocele and Myelic limited dorsal myeloschisis (MyeLDM) correspond to neural tube defects which lead to lifelong disabilities including lower extremity paralysis, sphincters deficiency, and cerebral complications (Chiari 2 malformation and hydrocephalus). It is demonstrated that fetal surgery repair of MMC with upper limit between the first thoracic vertebra (T1) and the first sacral vertebra (S1) improves motor and cerebral prognosis. Nowadays, this fetal surgery is performed either after maternal laparotomy and hysterotomy (open fetal surgery) or using fetoscopy. the investigators, at Trousseau Hospital (APHP, Paris), initiated an open fetal surgery of MMC program called PRIUM1 and 16 fetuses has been currently operated.

Fetoscopic repair of MMC is proposed by several international groups in order to prevent from maternal and obstetric morbidity related to the hysterotomy and improve the mother's obstetrical prognosis by allowing vaginal delivery. Results of fetoscopic MMC repair are very satisfying, both in terms of repair surgery efficacy and in terms of obstetrical prognosis. The research team believe that it is justified to propose this minimally invasive repair technique using fetoscopy, for represented by sacral MMC (level S1 and lower) as well as for intermediate forms between open and closed dysgraphisms, represented by MyeLDM. Indeed, these dysraphism are associated with the same cerebral complications than MMC with upper limit between T1 and S1 which could be corrected with prenatal repair. In addition, the spinal cord protection offered by prenatal surgery could prevent from the neuroepithelium destruction observed during pregnancy, with a potential motor benefit for the children.

The main objective of PRIUM 2 is to evaluate the success of fetoscopic surgical repair of sacral MMC or MyeLDM with a birth after 32 weeks of gestation and without severe perinatal morbidity and mortality.

The secondary objectives of PRIUM 2 are to evaluate the complications of pregnancy related to fetoscopic surgery as well as to evaluate the prenatal and postnatal evolution of the cerebral complications (Chiari 2 malformation and hydrocephalus) after fetoscopic repair surgery of the dysraphism (up to 12 months of age).

In this protocol, fetal sacral MMC/ MyeLDM repair surgery will be performed using gas fetoscopy before 26 weeks. After an exteriorization of the uterus through a laparotomy, humidified and warmed gas will be insufflated with low pressure (6 to 8mmHg mmHg). Fetoscopic repair surgery will be performed by a multidisciplinary team (maternal fetal medicine specialists, pediatric neurosurgeons, pediatric surgeons).

After discharge, patients will be followed weekly by a midwife and every two weeks by a referring obstetrician who will perform a clinical examination and a fetal ultrasound.A post procedure MRI will be performed 4 weeks after the surgery. If there is no obstetrical contraindication, vaginal delivery will be authorized.

The children will be followed according to the conventional management of children with dysraphisms and consultations at 8 weeks of life and 12 months of life will be scheduled at Trousseau Hospital, with the multidisciplinary team (pediatric neurosurgeons, physical medicine and rehabilitation specialists, pediatric orthopedic surgeons). During these two consultations, the children will have a complete clinical examination, a cerebral and spinal MRI and an ultrasound of the urinary tract.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria :

* Pregnant women age 18 years and older who are able to consent
* Singleton pregnancy before 26 weeks of gestation,
* Sacral MMC (upper level S1 or below) or MyeLDM diagnosed on ultrasound and MRI, 4. Absence of associated malformation apart from the anomalies usually observed in cases of open dysraphisms (i.e. feet malpositions, associated cerebral signs) or chromosomal anomaly if verification of the karyotype was desired by the couple
* Affiliated to health insurance, understanding and speaking French
* Written consent of the patient for the surgery and representatives of the parental authority for the postnatal follow-up of the child
* Patient who made the choice to continue the pregnancy

Exclusion Criteria:

* Abnormal angulation of the fetal spine,
* risk factors for prematurity: cervical length less < 15mm, history of late miscarriage before 22 weeks, pre-existing rupture of the membranes at inclusion,
* Placenta praevia,
* BMI greater than 35 kg / m2,
* Abnormality of the uterus: large fibroid, uterine malformation, history of uterine body surgery
* Maternal infection at risk of maternal-fetal transmission: HIV, HBV, HCV,
* Surgical or anesthetic contraindication.
* Participation in another interventional research protocol,
* Patients under legal protection (guardianship, curatorship).
* Allergies to drugs used in the research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-11-24 (Actual); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
Ability to perform fetoscopic sacral MMC/MyeLDM repair without severe perinatal morbidity and mortality | From time of surgery to 8 weeks of life (up to 28 weeks)
  Successful complete closure of the defect using the fetoscopic technique AND birth after 32 weeks without severe perinatal morbidity and mortality including grade III-IV intra ventricular hemorrhage, severe, cerebral parenchyma hemorrhage, periventricular leukomalacia, grade III ulcero-necrotizing enterocolitis, severe bronchodysplasia)

SECONDARY OUTCOMES:
Adverse Maternal outcome | during the surgery
  diagnosis of maternal gas embolism, hemorrhage, thromboembolic complication, death
Maternal obstetric outcome as evidenced by preterm labor leading to delivery at less than 37 weeks of gestation | From time of surgery until 37 weeks of gestation
  Preterm labor occuring at any time from surgery leading to delivery before 37 weeks of gestation
Maternal obstetric outcome as evidenced by preterm premature rupture of membranes | From time of surgery until 37 weeks of gestation
  Preterm premature rupture of membranes occuring at any time from surgery until 37 weeks of gestation
Maternal obstetric outcome as evidenced by chorioamnionitis | From time of surgery until 37 weeks of gestation
  chorioamnionitis occuring at any time from surgery until 37 weeks of gestation
Maternal obstetric outcome as evidenced by antenatal betamethasone treatment | From time of surgery until 34 weeks of gestation
  indication for a betamethasone course occuring at any time from surgery until 34 weeks of gestation
Other Maternal obstetric outcome as evidenced by hypertensive disorders, preeclampsia, gestational diabetes | From time of surgery until 37 weeks of gestation
  hypertensive disorders, preeclampsia, gestational diabetes occuring any time from surgery until 37 weeks of gestation
Prenatal evolution of brain abnormalities associated with open dysraphism, after fetoscopic repair | From time of surgery until birth
  Difference in the growth of the cephalic perimeter measured on an axial ultrasound section
Prenatal evolution of brain abnormalities associated with open dysraphism, after fetoscopic repair (1) | From time of surgery until birth
  Difference in measurement of the ventricles on an axial ultrasound section
Prenatal evolution of brain abnormalities associated with open dysraphism, after fetoscopic repair (2) | From time of surgery until birth
  Difference in the measurement of the large retro-cerebellar cistern on an axial section of the posterior fossa
Prenatal evolution of brain abnormalities associated with open dysraphism, after fetoscopic repair (3) | From time of surgery until birth
  Proportion of patients with reversal of hindbrain herniation (i.e. lower limit of the vermis located above the foramen magnum on ultrasound and/or fetal MRI)
Maternal obstetric outcome as evidenced by gestational age at delivery (1) | From time of surgery until delivery
  Gestational age of delivery regardless of indication
Maternal obstetric outcome as evidenced by gestational age at delivery (2) | From time of surgery until delivery
  Proportion of deliveries before 37 weeks of gestation
Maternal obstetric outcome as evidenced by the ability to deliver vaginally | From time of surgery until delivery
  Mode of delivery - either vaginal or cesarean section
Proportion of postpartum hemorrhages | From time of surgery until delivery
  Maternal obstetric outcome as evidenced by postpartum hemorrhage Proportion of postpartum hemorrhages defined by blood loss of more than 500mL for vaginal delivery, and 800mL for cesarean delivery
Need for maternal transfusion (number of blood cells transfused) | From time of surgery until delivery
  Maternal obstetric outcome as evidenced by postpartum hemorrhage Need for maternal transfusion (number of blood cells transfused)
Adverse neonatal outcome at birth (1) | at birth
  Normal or abnormal birth parameters at birth depending on the term
Adverse neonatal outcome at birth (2) | at birth
  Proportion of fetal asphyxia (arterial pH at the umbilical cord <7.00)
Adverse early childhood outcome as evidenced by need for a neurosurgical intervention | From the time of birth until 8 weeks of life
  need for one of the following neurosurgery
  * Type 1: Superficial skin recovery surgery due to scar dehiscence
  * Type 2: Need for surgical correction involving all aspects, without reopening the dura
  * Type 3: Need for complete surgical correction with repair of the dural plane
Postnatal evolution of brain abnormalities associated with open dysraphism | From the time of birth until 12 months of life
  Difference in the growth of the cephalic perimeter by measuring the cranial perimeter between birth and the age of 12 months
Postnatal evolution of brain abnormalities associated with open dysraphism (1) | From the time of birth until 12 months of life
  Difference in the measurement of the cerebral lateral ventricles measured during postnatal transfrontanellar ultrasound followed by cerebral MRI ,
Postnatal evolution of brain abnormalities associated with open dysraphism (2) | From the time of birth until 12 months of life
  Proportion of patients with reversal of hindbrain herniation (i.e. lower limit of the vermis located above the foramen magnum on cerebral MRI)
Postnatal evolution of brain abnormalities associated with open dysraphism (3) | From the time of birth until 12 months of life
  Proportion of patients requiring a cerebrospinal fluid shunt within the first 12 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Lucie GUILBAUD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service médecine foetale-Hôpital Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided